CLINICAL TRIAL: NCT07378189
Title: Opioid-free Anesthesia as an Alternative to General Anesthesia in Patients Undergoing Laparoscopic Peripheral Pancreatic Resection
Acronym: OFAPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, older asistent, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1072.6120.146.2025
Record Dates: First submitted 2025-12-25; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
Keywords: Pain; OFA; Opioid Free Anesthesia
MeSH Terms: conditions — Agnosia; Pain | interventions — Balanced Anesthesia; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balanced anesthesia with opioids (Active Comparator): Patients who will have pancreatic operation under balanced anesthesia including opioids
  Interventions: Drug: Balanced anesthesia with opioids
- Opioid Free Anesthesia (OFA) (Experimental): Patients who willl have pancreatic operation under Opioid Free anesthesia
  Interventions: Other: Opioid Free Anesthesia (OFA)

INTERVENTIONS:
Other: Opioid Free Anesthesia (OFA) — Patients who will have pancreatic operation under Opioid Free anesthesia
  Arms: Opioid Free Anesthesia (OFA)
Drug: Balanced anesthesia with opioids — Patients who will hav pancreatic operation under balanced anesthesia including opioids
  Arms: Balanced anesthesia with opioids

SUMMARY:
Opioid-free anesthesia is not associated with greater pain than opioid anesthesia and is associated with reduced postoperative pain.

DETAILED DESCRIPTION:
In our study, the investigators would like to compare the measurement of total oxycodone consumption in the postoperative period in both groups and whether the use of opioid-free anesthesia would reduce opioid consumption by 30%. The secondary objective will be to assess pain in both groups during the first 48 postoperative hours in patients undergoing pancreatic surgery. Patients would be randomly assigned to anesthesia with and without opioids at 1, 2, 6, 12, 24, and 48 hours after surgery. Other secondary objectives include assessing the incidence of postoperative nausea and vomiting (PONV), adverse drug reactions, particularly cardiac arrhythmias, and the impact on persistent postoperative pain. On day 7 after surgery, each patient will receive the QOR-15 questionnaire to assess quality of life and the PQA-10 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent to participate in the study
* Qualified for laparoscopic peripheral pancreatic resection
* Age 18-80 years
* ASA II and III

Exclusion Criteria:

* Patient refusal to participate in the study
* Inability to operate a PCA pump
* Lack of understanding of the NRS scale
* Hypersensitivity to anesthetics
* First- or second-degree heart block.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | up to 48 hours after surgery
  measurement of total oxycodone consumption in the postoperative period

SECONDARY OUTCOMES:
Pain assessment | at 1, 2, 6, 12, 24, and 48 hours after surgery
  Assessment of pain at 1, 2, 6, 12, 24, and 48 hours after surgery by NRS scale (0-10, 0 - no pain, 10 worst pain imaginable)
PONV | up to 48 h after surgery
  assessment of the occurrence of postoperative nausea and vomiting (PONV)
Quality Of Recovery | on the 7th day after surgery
  QOR-15 questionnaire to assess quality of life and PQA-10 questionnaire. The QOR-15 is a 15 items questionnaire which provides a valid and efficient evaluation of the postoperative quality of recovery.
  The QoR 15 score is a score of 15 items, each scored from 0 to 10. These items assess 5 dimensions of post-operative recovery: pain, physical comfort, functional autonomy, emotions and psychological support.
  These 15 items represent the quality of post-operative rehabilitation in its physical and mental dimensions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Intensive Interdisciplinary Care, Collegium Medicum, Jagiellonian University, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
ndividual participant data (IPD) will be shared contingent upon obtaining appropriate consent from the study participants. Data will be made available only in accordance with applicable ethical and regulatory requirements.